CLINICAL TRIAL: NCT01684150
Title: A Phase 1, Open-Label, Dose-Escalation & Expanded Cohort, Continuous IV Infusion, Multi-center Study of the Safety, Tolerability,PK & PD of EPZ-5676 in Treatment Relapsed/Refractory Patients With Leukemias Involving Translocation of the MLL Gene at 11q23 or Advanced Hematologic Malignancies
Brief Title: A Phase 1, Open-Label, Dose-Escalation & Expanded Cohort, Continuous IV Infusion, Multi-center Study of the Safety, Tolerability,PK & PD of EPZ-5676 in Treatment Relapsed/Refractory Patients With Leukemias Involving
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPZ-5676-12-001; 2013-002355-15 (EudraCT Number)
Record Dates: First submitted 2012-09-06; First posted 2012-09-12 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Disorders
Keywords: Leukemia; Advanced hematologic malignancies; Epizyme; Phase 1; Mixed Lineage Leukemia (MLL)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia | interventions — EPZ-5676

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPZ-5676 Extension cohort (Experimental)
  Interventions: Drug: EPZ-5676

INTERVENTIONS:
Drug: EPZ-5676 — MLL-r and MLL-PTD 28-day continuous IV infusion of each 28-day cycle. Number of cycles: until disease progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to determine the safe dose of EPZ-5676, to evaluate the safety of EPZ-5676 in patients with advanced hematologic malignancies, and to conduct a preliminary assessment of the anti-leukemia activity of EPZ-5676 in patients with acute leukemias bearing rearrangements of the MLL gene.

Currently this study is in the MLL-r restricted/expansion phase and is only enrolling patients with rearrangements involving the MLL gene, including 11q23 or partial tandem duplications (PTD).

DETAILED DESCRIPTION:
A subset of patients with acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL) harbor rearrangements of the MLL gene, which are detected either by cytogenetic or fluorescent in situ hybridization evaluation at the time of diagnosis. A protein called DOT1L plays an important role in the malignant process in these leukemias. EPZ-5676 is a molecule that blocks the activity of DOT1L, and is therefore being evaluated in the treatment of patients with MLL-rearranged leukemias.

The dose escalation portion has been completed. Currently this study is in the expansion phase and patients with MLL-r and MLL-PTD will receive EPZ-5676 as a 28-day continuous intravenous infusion (CIV).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years.
2. Patients with relapsed /refractory AML, ALL, or MLL with rearrangement of the MLL gene, including 11q23 or PTD, are eligible for the expanded cohort:

   * At least one prior therapy;
   * Refractory disease on most recent therapy, or disease recurrence following remission on most recent therapy;
   * Received and failed all known effective therapies for their disease;
   * Not a candidate for allogeneic stem cell transplantation
   * > 10% blasts or biopsy-documented leukemia cutis or myeloid sarcoma.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Patients must have the following clinical laboratory values:

   * Serum creatinine ≤2 mg/dL or creatinine clearance > 60 mL/minute;
   * Total bilirubin ≤2.0 times the ULN for the institution, unless considered due to Gilbert's syndrome;
   * ALT or AST ≤ twice the upper limit of normal (ULN), unless considered due to organ leukemic involvement;
   * Absolute neutrophil count ≥1,000/µL (unless due to documented leukemic involvement of the bone marrow at the time of study entry)
   * Platelets ≥100,000/µL (unless due to documented leukemic involvement of the bone marrow at the time of study entry).
   * PT or aPTT < 1.5 times the ULN
5. Able and willing to give written informed consent.
6. Life expectancy of at least 3 months

Exclusion Criteria:

1. Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
2. Active heart disease
3. Receiving any other standard treatment for their hematologic malignancy.
4. Receiving strong CYP3A4 inhibitors/ inducers.
5. Known history of cerebrovascular accident in the past 6 months.
6. Known bleeding diathesis.
7. Known, active (symptomatic) involvement of the central nervous system by leukemia.
8. On immunosuppressive therapy.
9. Known active infection.
10. Pregnant or nursing females.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of EPZ-5676 as determined by incidence of protocol-specified dose-limiting adverse events. | up to 12 months
  The MTD is defined as the dose level below in which >1 patient out of 3 or >2 patients out of 6 experience dose-limiting adverse events (as defined by the protocol).

SECONDARY OUTCOMES:
Pharmacokinetic profile of EPZ-5676 | up to 24 months
  analysis of Cmax, AUC and steady state concentration
The incidence of adverse events in patients treated with EPZ-5676 | up to 24 months
  Evaluation of adverse events, vital signs, physical examination, 12-lead ECG, and laboratory assessments
Anti-leukemic activity of EPZ-5676 in patients with acute leukemia harboring a MLL-rearrangement | up to 24 months
  Evaluation of response by standard criteria for AML or ALL
Effects of EPZ-5676 on histone H3K79 methylation in peripheral blood mononuclear cells (PBMC). | up to 24 months
Effects of EPZ-5676 on histone H3K79 methylation in leukemia cells | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Jesus Berdeja, MD, Principal Investigator — SCRI Development Innovations, LLC; David A Rizzieri, MD, Principal Investigator — Duke University; Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center; Jessica Altman, MD, Principal Investigator — Northwestern University; Raoul Tibes, MD, Principal Investigator — Mayo Clinic Scottsdale-Phoenix; Mojca Jongen-Lavrencic, MD, Principal Investigator — Erasmus Medical Center; Hartmut Döhner, MD, Principal Investigator — Universitätsklinikum Ulm; Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- United States (6):
  - Mayo Clinic Scottsdale-Phoenix, Scottsdale, Arizona
  - Northwestern University, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT MD Anderson Cancer, Houston, Texas
- Universitätsklinikum Ulm, Ulm, Germany
- Erasmus University Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Stein EM, Garcia-Manero G, Rizzieri DA, Tibes R, Berdeja JG, Savona MR, Jongen-Lavrenic M, Altman JK, Thomson B, Blakemore SJ, Daigle SR, Waters NJ, Suttle AB, Clawson A, Pollock R, Krivtsov A, Armstrong SA, DiMartino J, Hedrick E, Lowenberg B, Tallman MS. The DOT1L inhibitor pinometostat reduces H3K79 methylation and has modest clinical activity in adult acute leukemia. Blood. 2018 Jun 14;131(24):2661-2669. doi: 10.1182/blood-2017-12-818948. Epub 2018 May 3. PMID 29724899